CLINICAL TRIAL: NCT04922528
Title: Evaluate the Efficacy of ICG Fluorescent Cholangiography for Visualization of Extrahepatic Biliary Anatomy in Emergency Cholecystectomy: A Single-Center, Randomized, Controlled, Parallel-Group Study
Brief Title: Visualization of the Extrahepatic biliaRy Tree Trial
Acronym: VERT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Philip Dawe, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H21-01375
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Cholecystitis, Acute; Acute Cholangitis; Gallstone Pancreatitis; Choledocholithiasis; Cholecystolithiasis; Gallbladder Diseases; Biliary Tract Diseases; Digestive System Disease; Calculi; Pathological Conditions, Anatomical
Keywords: Cholangiography; Indocyanine green; ICG; Fluorescent cholangiography; Biliary Anatomy
MeSH Terms: conditions — Cholecystitis, Acute; Choledocholithiasis; Cholecystolithiasis; Gallbladder Diseases; Biliary Tract Diseases; Digestive System Diseases; Calculi; Pathological Conditions, Anatomical | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: The intervention and comparator arms will be ran in parallel, with a block randomization sequence determining the participants allocations.
Who Masked: Participant
Masking Description: Due to the procedural nature of the intervention, we have chosen to run this trial single-blinding, with only the participant being masked to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Near-Infrared Fluorescence Cholangiography (Experimental): Standard laparoscopic cholecystectomy completed with a combination of white light imaging and near-Infrared fluorescence cholangiography after administering 5 mg of a 25 mg/10 mL solution of indocyanine green (ICG) intravenously prior to the operation
  Interventions: Procedure: Laparoscopic Cholecystectomy with Fluorescent Cholangiography; Procedure: Laparoscopic Cholecystectomy with White Light Imaging
- White Light Imaging (Active Comparator): Standard laparoscopic cholecystectomy completed with only standard white light imaging only
  Interventions: Procedure: Laparoscopic Cholecystectomy with White Light Imaging

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy with Fluorescent Cholangiography — Indocyanine green is a fluorophore molecule which is metabolized by the liver and excreted exclusively through the biliary system. Intra-operatively, near-infared imaging via the laparoscope will be used to visualize the biliary anatomy in the intervention arm, as an adjunct to standard of care white-light imaging.
  Arms: Near-Infrared Fluorescence Cholangiography
Procedure: Laparoscopic Cholecystectomy with White Light Imaging — As per the current standard of care, patients undergoing laparoscopic cholecystectomies will have it completed using white light imaging through the laparoscope.

SUMMARY:
This study is a prospective randomized controlled trial evaluating the use of a fluorescent dye, indocyanine green (ICG), in the identification of important bile duct anatomy during emergent same-admission cholecystectomy. Participants will be randomized into either the control arm, which uses the standard of care white light during laparoscopy or the intervention arm, which will use ICG fluorescent cholangiography as an adjunct to white light to visualize the biliary anatomy. The investigators hypothesize that the use of fluorescent cholangiography will increase the rates of identification of important biliary anatomy during laparoscopic cholecystectomy. The effectiveness, feasibility, and safety will be compared between the two groups using a post-operative survey form the surgeons will complete prior to exiting the operating room.

DETAILED DESCRIPTION:
Near-infrared fluorescent imaging techniques have shown promise in aiding to delineate and visualize extrahepatic biliary structures. Indocyanine green (ICG) is a water-soluble fluorescent dye that has been shown to improve visualization of biliary anatomy under fluorescent cholangiography. The standard of care for many acute biliary disease conditions, such as acute cholecystitis, remains early laparoscopic cholecystectomy. Even though real-time fluorescent cholangiography using ICG has the potential to enhance the visualization of biliary structures and anatomy, and therefore reduce the risk for bile duct injury, the majority of the studies published to date exclude acute biliary disease patients. The pathophysiology of acute biliary disease processes is associated with inflammation and adhesions that increase the challenge of achieving a critical view of safety. The investigators propose that using ICG and fluorescent cholangiography near-infrared imaging techniques as an adjunct in acute care laparoscopic cholecystectomies has the potential to help mitigate the increased risk of bile duct injury by increasing extrahepatic biliary structure detection and surgeon confidence.

Eligible patients will be identified through their initial clinical evaluation, which will be verified by the patient's primary surgeon. If and once a patient has been confirmed as eligible, the surgeon or designate will introduce the clinical trial design in detail. If after being introduced to the study and having had the opportunity to ask questions, the patient is willing to participate, the patient will be asked to review and sign the informed consent document.

Upon entry into the clinical trial, the allocation sequence will be generated using a block randomization schema with computer-generated random numbers in a 1:1 ratio, with block sizes of 4 by a co-investigator with no clinical involvement in the trial. The same co-investigator will prepare sequentially numbered, opaque, sealed and stapled envelopes and stored them in a locked cabinet in the operating room control desk. Each envelope contained instructions for the arm the participant had been randomly assigned to, either treatment (ICG cholangiography) or control (standard white light only) arms. After the research team member has obtained the participant's consent, the surgeon or designates will obtain the next consecutively numbered envelope and proceed to open it after the patient is anesthetized and prior to beginning the surgery.

The patient will be blinded to the result of the randomization until after surgery as the envelope will be opened only after the patient has received their general anesthetic. No blinding of the surgical team, research team members or outcomes assessors will be used in this study given the procedural nature and acute condition of the patients included.

ELIGIBILITY:
Inclusion Criteria:

* Admission or consultation by the Acute Care Surgery (ACS) service
* Diagnosis of acute biliary disease requiring index laparoscopic cholecystectomy
* Diagnoses of acute cholangitis, choledocholithiasis, and gall stone pancreatitis may be included. However, they must have cleared ducts confirmed via endoscopic ultrasound, ultrasound, ERCP, and/or laboratory investigations.
* Ability to understand and follow study procedures and protocols, and provide signed informed consent.

Exclusion Criteria:

* Female patients who are pregnant or currently breastfeeding
* Known pre-existing liver disease, including cirrhosis
* Known allergy to iodine or shellfish
* Known allergy to indocyanine green (ICG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of extrahepatic biliary structures | Intraoperatively
  The extrahepatic biliary structures which we will be assessing the identification of include: Cystic Duct (CD), Right Hepatic Duct (RHD), Common Hepatic Duct (CHD), Common Bile Duct (CBD), Cystic Duct - Gall Bladder junction (CD-GB), and Cystic Duct - Common Bile Duct junction (CD-CBD).

SECONDARY OUTCOMES:
Operative success | Intraoperatively
  Rates of laparoscopic subtotal cholecystectomy and laparoscopic cholecystostomy tube placement.
Rates of conversion | Intraoperatively
  Rate of conversion to open cholecystectomy.
Operative time | Intraoperatively
  From the time of opening the skin to the time of closure.
Surgeon satisfaction | Through participant discharge, an average of 1 week
  Operating surgeons satisfaction (as rated by post-procedural survey) with the utility and feasibility of the modality.

OTHER OUTCOMES:
Adverse events | Through participant discharge, an average of 1 week
  Any adverse events associated with the administration or use of ICG fluorescent cholangiography
Procedural complications | Through participant discharge, an average of 1 week
  Any complications associated with the cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philip Dawe, CD MD FRCSC, Principal Investigator — Clinical Assistant Professor
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zroback C, Chow G, Meneghetti A, Warnock G, Meloche M, Chiu CJ, Panton ON. Fluorescent cholangiography in laparoscopic cholecystectomy: the initial Canadian experience. Am J Surg. 2016 May;211(5):933-7. doi: 10.1016/j.amjsurg.2016.01.013. Epub 2016 Feb 23. PMID 27151917
- [Background] Bleszynski MS, DeGirolamo KM, Meneghetti AT, Chiu CJ, Panton ON. Fluorescent Cholangiography in Laparoscopic Cholecystectomy: An Updated Canadian Experience. Surg Innov. 2020 Feb;27(1):38-43. doi: 10.1177/1553350619885792. Epub 2019 Nov 19. PMID 31744398